CLINICAL TRIAL: NCT06532578
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Multicenter Trial to Evaluate the Safety and Efficacy of CPX101 in Overweight and Obese Subjects Without Diabetes Mellitus
Brief Title: Evaluate the Safety and Efficacy of CPX101 in Overweight and Obese Subjects Without Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Chia Tai Innovative Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPX101-Ⅱ-01
Record Dates: First submitted 2024-07-18; First posted 2024-08-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Biological: CPX101 or placebo 120mg Q2W
- Cohort 2 (Experimental)
  Interventions: Biological: CPX101 or placebo 160mg Q4W
- Cohort 3 (Experimental)
  Interventions: Biological: CPX101 or placebo 160mg Q2W
- Cohort 4 (Experimental)
  Interventions: Biological: CPX101 or placebo 240mg Q4W; Biological: CPX101 or placebo 360mg Q4W
- Cohort 5 (Experimental)
  Interventions: Biological: CPX101 or placebo 240mg Q2W; Biological: CPX101 or placebo 360mg Q2W

INTERVENTIONS:
Biological: CPX101 or placebo 120mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: Cohort 1
Biological: CPX101 or placebo 160mg Q4W — Subcutaneous injection of CPX101 or placebo
  Arms: Cohort 2
Biological: CPX101 or placebo 160mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: Cohort 3
Biological: CPX101 or placebo 240mg Q4W — Subcutaneous injection of CPX101 or placebo
  Arms: Cohort 4
Biological: CPX101 or placebo 240mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: Cohort 5
Biological: CPX101 or placebo 360mg Q2W — CPX101 or placebo 360mg Q2W
  Arms: Cohort 5
Biological: CPX101 or placebo 360mg Q4W — CPX101 or placebo 360mg Q4W
  Arms: Cohort 4

SUMMARY:
The study is designed to evaluate the preliminary efficacy, safety, population PK profile, and immunogenicity of CPX101 in subjects with obesity or overweight with weight related comorbidities but without diabetes mellitus.

DETAILED DESCRIPTION:
240 subjects who meet the eligibility criteria will be randomized to 5 cohorts in a 2:3:3:2:2 ratio (CPX101 120mg Q2W, CPX101 160mg Q4W, CPX101 160mg Q2W, CPX101 240mg Q4W, CPX101 240mg Q2W).Participants in each cohort will be randomized in a 3:1 ratio to receive either CPX101 or placebo. The study consists of a 3-week screening period, a 24-week treatment period, and a 12-week safety follow-up period.Dose-titration will be adopted within each cohort to improve GI tolerability.

ELIGIBILITY:
5.1 Inclusion Criteria Subjects who are eligible for the study must meet all of the following core inclusion criteria.

1. Provide signed informed consent.
2. Males or females aged 18-75 years (inclusive) at the time of signing the informed consent form (ICF).
3. Body mass index (BMI) ≥ 30 kg/m2, or 27≤BMI<30 kg/m2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): pre-diabetes, hypertension, dyslipidaemia, obstructive sleep apnoea, ischemic cardiovascular disease, or concomitant weight-bearing joint pain.
4. Body weight is stable during the 3-month period prior to screening, and any weight change is less than 5%.
5. In the investigator's opinion, are capable and willing to follow the study procedure of the study, including but not limited to: follow lifestyle advice (for example, dietary restrictions and exercise plan), maintain a study diary, and complete required questionnaires.
6. At least one self-reported unsuccessful weight loss attempt per investigator judgement.
7. Satisfy the following:

   a) For female subjects: i. Female subjects with childbearing potential: Serum pregnancy test result at screening must be negative, and must agree to use at least one of the effective contraceptive methods (refer to appendix 4) from the time of signing the ICF until 12 weeks after the last dose of study drug. If a female subject decides to use any one of user-dependent contraceptive method (refer to Appendix 4), then a second method of contraceptive barrier is required.

ii. Female subjects with non-childbearing potential: Postmenopausal for at least 12 months, or documented surgically sterile (e.g. hysterectomy, with or without bilateral salpingectomy and bilateral oophorectomy). Females who have only had tubal ligation or other birth control operations are NOT included.

b) For male subjects: all male subjects should refrain from sperm donation from the time of signing the ICF until 12 weeks after the last dose of study drug. If engaged in sexual relations with a female of child-bearing potential, subjects must use condoms plus 1 additional highly effective (refer to appendix 4) method of contraception during intercourse from the time of signing the ICF until 12 weeks after the last dose of study drug.

5.2 Exclusion Criteria

Subjects are excluded from the trial if any of the following criteria apply:

Glycaemia-related:

1. HbA1c ≥6.5% at screening or diagnosed with type 1 or type 2 diabetes mellitus.
2. Treatment with glucose-lowering agent(s) within 90 days before screening.
3. There are severe hypoglycemic events of unknown cause (needing help from others to recover) from 90 days before screening to randomization, or frequent hypoglycemia such as 3 or more hypoglycemic events (blood glucose ≤ 2.8 mmol/L) or hypoglycemia-related symptoms within 30 days before screening.

   Obesity-related:
4. Treatment with GLP-1 receptor (GLP-1R) agonists or GLP-1R/GCGR agonists or GIPR/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists, or any other medication for the indication of obesity within 3 months before screening.
5. Previous or planned (during the trial period) obesity treatment with surgery or a weight loss device excluding liposuction and/or abdominoplasty, if performed > 1 year before screening.
6. Use of drugs with an impact on body weight within 3 months before screening based on investigator's opinion.
7. Presence of any clinically significant endocrine disorders (e.g., uncontrolled hyperthyroidism, or hypothyroidism, acromegaly, Cushing syndrome, etc.), which makes the participant unsuitable for the study, as the discretion of the investigator.

   Mental health:
8. Have a history of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 years before screening.
9. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15 at screening.
10. A lifetime history of a suicidal attempt, or suicidal behavior within 30 days before screening.
11. Suicidal ideation corresponding to Category 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 30 days before screening.

    General safety:
12. History of acute or chronic pancreatitis, history of symptomatic gallbladder disease (participants can be enrolled if gallbladder disease has been resolved by cholecystecomy), history of pancreatic injury, and other high-risk factors that may lead to pancreatitis.
13. History of clinically significant gastric emptying abnormalities (e.g., gastric outlet obstruction), serious chronic gastrointestinal disorders (e.g., active ulcer within 6 months before screening), long-term use of drugs with a direct impact on gastrointestinal motility, or gastrointestinal surgery (excluding endoscopic resection of gastrointestinal polyps, and appendicectomy).
14. Personal or family history of multiple endocrine neoplasia (MEN) syndrome type 2 or medullary thyroid carcinoma (MTC).
15. History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer, in situ carcinomas of the cervix, in situ prostate cancer and in situ melanoma are allowed.
16. History of major cardiovascular and cerebrovascular diseases within 6 months before screening, defined as:

    1. History of myocardial infarction, coronary angioplasty or bypass graft, valvular heart disease or valve repair, clinically significant arrhythmia, unstable angina, transient ischemic attack, or cerebrovascular accident;
    2. New York Heart Association (NYHA) class III or IV congestive cardiac failure;
    3. Or presence of abnormal ECG manifestations (excluding stable coronary heart disease) that may affect the safety judgment of the study or require medical intervention, at the discretion of the investigator.
17. Occurrence of serious trauma, serious infection, or surgery within 30 days before screening, which makes the participant unsuitable for the study, at the discretion of the investigator.
18. Known or suspected hypersensitivity to trial product(s) or related products.
19. Known or suspected abuse of alcohol (that is, alcohol consumption >14 units/week for women and >21 units/week for men) or recreational drugs.
20. Previous participation in this trial. Participation is defined as signed informed consent.
21. Participation in another clinical trial within 90 days before screening.
22. The physical examination or lab results at screening meet any of the following criteria:

    1. Blood pressure: systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg, or systolic blood pressure (SBP) ≤ 85 mmHg and/or diastolic blood pressure (DBP) ≤ 55 mmHg, or addition/change or dose adjustment of antihypertensive drugs within 4 weeks before screening;
    2. Liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 × the upper limit of normal (ULN); or total bilirubin > 1.5 × ULN; or alkaline phosphatase (ALP) > 1.5 × ULN;
    3. Pancreatic function: amylase and/or lipase > 1.5 × ULN;
    4. Renal function: renal impairment measured as estimated Glomerular Filtration Rate (eGFR, calculated by 2021 CKD-EPI) 30 ml/min/1.73 m2 at screening;
    5. Anemia of any cause, defined as hemoglobin < 120 g/L (male) or < 110 g/L (female) at screening;
    6. Fasting triglyceride > 5.7 mmol/L, or addition/change or dose adjustment of lipid-lowering drugs within 4 weeks before screening;
    7. Calcitonin ≥ 20 ng/L;
    8. Positive for any of the following: hepatitis B virus DNA (HBV DNA) ≥500IU/mL, hepatitis C virus RNA (HCV RNA) positive (≥the lowest value that can be tested), and human immunodeficiency virus (HIV) antibody.
23. Surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the investigator.
24. Female who is pregnant, breast-feeding or intends to become pregnant.
25. Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardise the subject's safety or compliance with the protocol.

The criteria will be assessed at the investigator's discretion unless otherwise stated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of CPX101 in body weight loss in Kg | Up to 24 weeks after administration
  To evaluate the efficacy of CPX101 in body weight loss by dose levels after 24 weeks of multiple subcutaneous injections in overweight and obese subjects without diabetes mellitus.

SECONDARY OUTCOMES:
Other efficacy parameters of CPX101(Waist circumference in centimeters) | Up to 24 weeks after administration
  To evaluate the efficacy of waist circumference of CPX101 by dose levels after 24 weeks of multiple subcutaneous injections in overweight and obese subjects without diabetes mellitus
Other efficacy parameters of CPX101(BMI) | Up to 24 weeks after administration
  BMI = wight (kg)/(height[m])^2 ;To evaluate BMI of CPX101 by dose levels after 24 weeks of multiple subcutaneous injections in overweight and abese subjects without diabetes mellitus.
Incidence of AE/SAE | Up to 36 weeks
  The safety of CPX101
The plasma concentration of CPX101 | Up to 24 weeks after administration
  Measurement of the plasma concentration of CPX101 in serum after multiple subcutaneous injections in overweight and obese subjects without diabetes mellitus.
Immunogenicity of CPX101 | Up to 24 weeks after administration
  Measurement of the anti-CPX101 antibody in serum after multiple subcutaneous injections in overweight and obese subjects without diabetes mellitus.

OTHER OUTCOMES:
Efficacy of CPX101 in body weight loss in Kg | At week 36
  To evaluate the efficacy of CPX101 in body weight loss at week 36 in overweight and obese subjects without diabetes mellitus

CONTACTS AND LOCATIONS:
Locations (1):
- Paratus Clinical Research, Chatswood, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No